CLINICAL TRIAL: NCT03580200
Title: Effects of Deep Trigger Point Dry Needling on Strength Measurements of the Gluteus Medius Musculature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emily Slaven, PT, PhD (Other)
Collaborators: Mount St Joseph University (Unknown)
Responsible Party: Sponsor-Investigator, Emily Slaven, PT, PhD, Professor, University of Indianapolis
Organization: University of Indianapolis (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0897-MSJU
Record Dates: First submitted 2018-05-25; First posted 2018-07-09 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Trigger Point; Muscle Weakness
Keywords: Latent Trigger Point; Myofascial Trigger Point; Trigger Point Dry Needling; Deep Dry Needling; Muscle Strength; Gluteus Medius
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study utilizing a pretest-posttest randomized control design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Side (Experimental): Each participant is to be randomly assigned an intervention side (side of the body that will receive trigger point dry needling) and a control side (side of the body that will not receive trigger point dry needling).
  Interventions: Other: Trigger Point Dry Needling
- Control Side (No Intervention): Each participant is to be randomly assigned an intervention side (side of the body that will receive trigger point dry needling) and a control side (side of the body that will not receive trigger point dry needling).

INTERVENTIONS:
Other: Trigger Point Dry Needling — For the purposes of this study, the term trigger point dry needling will be used to describe deep dry needling of muscle tissue. The goal of trigger point dry needling is to eliminate myofascial trigger points within muscle tissue, thereby reducing pain as well as improving motor control and function (Caramagno et al., 2015; Dommerholt et al., 2006; Shah et al., 2015). Trigger point dry needling utilizes a solid filiform needle and focuses on the penetration of a palpable myofascial trigger point at various depths. The needle is then manipulated within the tissue in an attempt to elicit a localized twitch response. Once the localized twitch response has ended, the needle is removed and another myofascial trigger point is located.
  Other Names: Deep Dry Needling
  Arms: Intervention Side

SUMMARY:
The purpose of this study will be to assess the effect that the application of deep trigger point dry needling to latent trigger points has on strength measurements. Specifically, the effect of deep trigger point dry needling on the strength measurements of the gluteus medius musculature immediately following intervention will be investigated. The author hypothesizes that there will be a significant difference in strength measurements of the gluteus medius musculature between the intervention and controls sides as well as within the intervention and control sides prior to and immediately following the application of deep trigger point dry needling. It is the authors' intention that clinicians may be able to apply the results of this study to generate a safe and effective treatment plan that can reduce the risk for trunk and lower extremity injuries within their patient population by reducing the number of latent trigger points within muscle tissue.

ELIGIBILITY:
Inclusion Criteria:

Males and females will be included in the study if they are between the ages of 18 and 50 years and are currently asymptomatic at the time of screening and data collection. Asymptomatic will be defined as individuals who are currently experiencing no pain in their lumbar spine, sacroiliac region, pelvis, or bilateral lower extremities while at rest or with activity.

Exclusion Criteria:

Participants will be excluded from the study if they have one of the following:

* Currently pregnant as self-reported by the participant
* Pain intensity greater than 0 out of 10 on the visual analogue scale in the lumbar spine, sacroiliac region, pelvis, and bilateral lower extremities at rest or with activity
* Positive Flexion Adduction Internal Rotation (FADIR) test on either the left or right hip. If the individual experiences a reproduction of his or her pain response with the FADIR test, which is overpressure into hip flexion, adduction, and internal rotation, he or she will be excluded from participation in the study
* Present with signs and symptoms consistent with hip osteoarthritis during clinical screening using the criteria proposed Altman et al. (1991) on either the left or right hip. Criteria is as follows: If an individual presents with pain in the hip joint with hip internal rotation that is measured to be less than 15 degrees as well as hip flexion that is measured to be less than or equal to 115 degrees, they will be excluded from participation in the study.
* Diagnosed with a progressive neurological disorder that may affect the strength of their lower extremities, a chronic pain condition such as fibromyalgia or myofascial pain syndrome, a connective tissue disorder such as Ehlers-Danlos syndrome, or osteoarthritis of the hip joint
* History of hip dysplasia or Legg Calve Perthes disease

In order to continue within the study once the inclusion criteria has been met. Participants will be required to have at least 2 palpable latent trigger points in the gluteus medius muscle on the intervention sides. Individuals that do not have greater than 2 latent trigger points on the intervention side will not be allowed to continue with the study. Data already collected for these participants will be destroyed.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
The Degree of Change in the Strength of the Gluteus Medius Musculature Measured by a Hand Held Dynamometer | Strength measurements of the gluteus medius will be recorded prior to and immediately following the application of trigger point dry needling for both the control & intervention sides to determine if a significant change in muscle strength has occurred.
  Strength of the gluteus medius musculature will be assessed for both the control and intervention sides. Strength of the gluteus medius muscle will be assessed using a hand held dynamometer which will measure peak force in kilograms. A maximal volitional isometric contraction break test will be used with the hip in two separate positions. A total of three measurements will be taken for each position and these measurements will be averaged for the hand held dynamometer readings. Both within group and between group differences in strength measurements will be compared for significance.
The Degree of Change in the Strength of the Gluteus Medius Musculature Measured by Surface Electromyography | Strength measurements of the gluteus medius will be recorded prior to & immediately following the application of trigger point dry needling for both the control and intervention sides to determine if a significant change in muscle strength has occurred.
  Strength of the gluteus medius musculature will be assessed for both the control and intervention sides. Strength of the gluteus medius muscle will be assessed using surface electromyography readings which will measure peak muscle contraction in millivolts. A maximal volitional isometric contraction break test will be used with the hip in two separate positions. A total of three measurements will be taken for each position and these measurements will be averaged for the surface electromyography readings. Both within group and between group differences in strength measurements will be compared for significance.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Slaven, PT, PhD, OCS, Principal Investigator — University of Indianapolis
Locations (1):
- Mount St Joseph Univeristy, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altman R, Alarcon G, Appelrouth D, Bloch D, Borenstein D, Brandt K, Brown C, Cooke TD, Daniel W, Feldman D, et al. The American College of Rheumatology criteria for the classification and reporting of osteoarthritis of the hip. Arthritis Rheum. 1991 May;34(5):505-14. doi: 10.1002/art.1780340502. PMID 2025304
- [Background] Caramagno J, Adrian L, Mueller L, Purl J. Analysis of competencies for dry needling by physical therapists: Final report. Federation of State Boards of Physical Therapy. https://www.apta.org/uploadedFiles/APTAorg/Advocacy/State/Issues/Dry_Needling/AnalysisCompetenciesforDryNeedlingbyPT.pdf. Published July 2015. Accessed May 21, 2018.
- [Background] Shah JP, Thaker N, Heimur J, Aredo JV, Sikdar S, Gerber L. Myofascial Trigger Points Then and Now: A Historical and Scientific Perspective. PM R. 2015 Jul;7(7):746-761. doi: 10.1016/j.pmrj.2015.01.024. Epub 2015 Feb 24. PMID 25724849
- [Background] Dommerholt J, Carel B, Franssen J. Myofascial trigger points: An evidence-informed review. Journal of Manual & Manipulative Therapy14(4): 203-221, 2006.